CLINICAL TRIAL: NCT00525005
Title: A Phase II Study of Docetaxel, Oxaliplatin and S-1 (DOS) in Patients With Advanced Gastric Cancer
Brief Title: Docetaxel, Oxaliplatin and S-1 (DOS) for Advanced Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hallym University Medical Center (Other)
Collaborators: Asan Medical Center (Other); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMC-HO-GI-0701
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasm; Docetaxel; Oxaliplatin; S-1
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Oxaliplatin; S 1 (combination); titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DOS (Docetaxel, Oxaliplatin and S-1) (Experimental): Docetaxel 52.5mg/m2 IV on D1 (diluted in 250 ml of normal saline over a 1 hour of each cycle before oxaliplatin) Oxaliplatin 105mg/m2 IV on D1 (diluted in 250 ml of 5% DW for 2 hours) S-1 80mg/m2/day on D1-14 (2 weeks of treatment followed by a 1-week rest period)
  Interventions: Drug: DOS (Docetaxel, Oxaliplatin and S-1)

INTERVENTIONS:
Drug: DOS (Docetaxel, Oxaliplatin and S-1) — Docetaxel 52.5mg/m2 IV on D1 (diluted in 250 ml of normal saline over a 1 hour of each cycle before oxaliplatin) Oxaliplatin 105mg/m2 IV on D1 (diluted in 250 ml of 5% DW for 2 hours) S-1 80mg/m2/day on D1-14 (2 weeks of treatment followed by a 1-week rest period)
  Other Names: Taxotere; Eloxatin; TS-1

SUMMARY:
The purpose of this study is to determine the efficacy of combination of docetaxel, oxaliplatin, and S-1 (DOS) in the treatment of advanced gastric cancer.

DETAILED DESCRIPTION:
Docetaxel is an anti-microtubule agent. Docetaxel is an active agent for gastric cancer, with response rate (RR) of 20-24% as a single agent and RR of 37-40% as a combination therapy with 5-FU and/or cisplatin.

S-1 is a new oral dihydropyrimidine dehydrogenase (DPD) inhibitory fluoropyrimidine (DIF). In two late phase II studies of S-1 for advanced gastric cancer, RR was 45%, with very low (2%) incidence of grade 3 toxicity.

Recent phase I/II trial of the combination of docetaxel and S-1 in patients with advanced gastric cancer suggests that repeated 3-4 week cycles of S-1 60-80mg/m2 /day for 14 days combined with docetaxel 40-75mg/m2 is feasible.

Oxaliplatin, diaminocyclohexane-platinum, is an alkylating agent inhibiting DNA replication. Comparing to cisplatin or carboplatin, oxaliplatin appear to be more effective and has a more favorable toxicity profile. Phase II studies of the combination of docetaxel and oxaliplatin in patients with advanced gastric cancer suggests that docetaxel 60 or 75mg/m2 combined with oxaliplatin 130 or 80mg/m2 every 3 weeks is feasible.

Recent dose finding study of the combination of docetaxel, oxaliplatin and S-1 (DOS) in patients with advanced gastric cancer suggests that docetaxel 52.5mg/m2 on day 1 and oxaliplatin 105mg/m2 on day 1 combined with S-1 80mg/m2 on day1 to day 14 every 3 weeks is feasible.

Docetaxel, S-1 and oxaliplatin have distinct mechanisms of action and no overlapped key toxicities. Furthermore, fluoropyrimidine and docetaxel or oxaliplatin have shown synergism in vivo studies and in clinical trials. Based on these results, the combination of DOS is a reasonable candidate of new chemotherapeutic regimen for the advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric adenocarcinoma, initially diagnosed or recurred
* Unresectable, locally advanced or metastatic
* At least one uni-dimensional measurable lesion by RECIST criteria
* Age 18 to 70 years old
* ECOG performance status ≤2
* Estimated life expectancy ≥3 months
* Adequate bone marrow function (WBCs ≥4,000/µL or absolute neutrophil count ≥1,500/µL, platelets ≥100,000/µL),
* Adequate kidney function (creatinine <1.5 mg/dL)
* Adequate liver function (bilirubin ≤1.8 mg/dL, transaminase levels <2 times the upper normal limit
* Written informed consent

Exclusion Criteria:

* Other tumor type than adenocarcinoma
* Previous history of chemotherapy (exception: adjuvant chemotherapy)
* Presence of CNS metastasis, psychosis, or seizure
* Obvious bowel obstruction
* Evidence of serious gastrointestinal bleeding
* Peripheral neuropathy (NCI CTC >= Grade I)
* Past or concurrent history of neoplasm other than gastric adenocarcinoma, except for curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix uteri
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Other serious illness or medical conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
overall response rate | 2.5 years

SECONDARY OUTCOMES:
safety, progression-free survival, and overall survival | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dae Young Zang, MD, PhD, Principal Investigator — Hallym University Medical Center
Locations (2):
- South Korea (2):
  - Hallym University Medical Center, Anyang
  - Asan Medical Center, Seoul

REFERENCES:
- [Background] Yamaguchi K, Shimamura T, Hyodo I, Koizumi W, Doi T, Narahara H, Komatsu Y, Kato T, Saitoh S, Akiya T, Munakata M, Miyata Y, Maeda Y, Takiuchi H, Nakano S, Esaki T, Kinjo F, Sakata Y. Phase I/II study of docetaxel and S-1 in patients with advanced gastric cancer. Br J Cancer. 2006 Jun 19;94(12):1803-8. doi: 10.1038/sj.bjc.6603196. PMID 16773074
- [Background] Yoshida K, Ninomiya M, Takakura N, Hirabayashi N, Takiyama W, Sato Y, Todo S, Terashima M, Gotoh M, Sakamoto J, Nishiyama M. Phase II study of docetaxel and S-1 combination therapy for advanced or recurrent gastric cancer. Clin Cancer Res. 2006 Jun 1;12(11 Pt 1):3402-7. doi: 10.1158/1078-0432.CCR-05-2425. PMID 16740764
- [Background] Zang D, Song H, Kwon J, Jung J, Kim H, Kim J, Shin H, Park Y. Phase I/II trial with docetaxel and S-1 for patients with advanced or recurrent gastric cancer. Ann Oncol. 2006 Sep 29;17(S9):ix314, Abs:1097P
- [Background] Richards D, Wilfong L, Sborov M, McCollum D, Khan M, Boehm K, Zhan F. Phase II trial of docetaxel+oxaliplatin in advanced gastroesophageal and/or stomach cancer. 7th World Congr Gastrointest cancer. 2005: Abs: P-143
- [Background] Barone C, Basso M, Schinzari G, Pozzo C, Trigila N, D'Argento E, Quirino M, Astone A, Cassano A. Docetaxel and oxaliplatin combination in second-line treatment of patients with advanced gastric cancer. Gastric Cancer. 2007;10(2):104-11. doi: 10.1007/s10120-007-0415-x. Epub 2007 Jun 25. PMID 17577620
- [Background] Zang D, Yang D, Lee H, Lee B, Hwang S, Kim H, Song H, Jung J, Kim J, Kwon J. Phase I study of docetaxel, oxalipaltin and S-1 (DOS) for patients with advanced gastric cancer. Ann Oncol 2007 Sep 23; Abs:in press